CLINICAL TRIAL: NCT05307133
Title: Oxytocin Serum Variation Following Laparoscopic Sleeve Gastrectomy in Morbidly Obese Women
Brief Title: Oxytocin and Sleeve Gastrectomy
Acronym: BARIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-AOI-12
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre menopausal women undergoing sleeve gastreexctomy for morbid obesity (Other): After the indication for sleeve gastrectomy has been retained by the multidisciplinary committee eligible patients will be contacted and offered to participate in the BARIAXYTOCINE study. At the time of the first outpatient visit (V1), body densitometry and blood sample for estradiol, leptin and oxytocin will be done. Patients will undergo surgery within one month and 6 months after surgery they will undergo the same work-up (V2).
  Interventions: Other: Sleeve Gastreextomy

INTERVENTIONS:
Other: Sleeve Gastreextomy — The aim of the present study is to elucidate whether serum levels of oxytocin and sleeve gastrectomy induced weight loss are correlated in pre-menopausal morbidly obese women.

SUMMARY:
Morbid obesity has become a common condition and there is no effective drug that is able to induce a sustained weight loss. Currently bariatric surgery remains the only effective means that is able to lead to long term sustained weight loss. Oxytocin is a hormone secreted by the hypophysis that regulates negatively the adipogenesis and positively the osteogenesis. Oxytocin also regulates appetite and its role in weight loss in humans has not been investigated so far. The aim of the present study is to elucidate whether plasma levels of oxytocin and sleeve gastrectomy induced weight loss are correlated in pre-menopausal morbidly obese women.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-65, pre-menopausal,
* able to read and understand the written informed consent,
* with a BMI > 40 or 35
* with at least one obesity linked comorbidity among blood hypertension,
* type 2 diabetes,
* sleep apnea syndrome,
* invalidating arthritis,
* indication for sleeve gastrectomy
* accepted by the multidisciplinary committee and the CPAM (local health care system agency),
* affiliation to the Fre,nch health care system,
* signature of the informed consent.

Exclusion Criteria:

* Post-menopausal women,
* any other bariatric procedure that sleeve gastrectomy, history of any other bariatric procedure,
* pregnancy,
* age less than 18 years under, under guardianship
* Patients undergoing any other procedure that the planned sleeve gastrectomy or undergoing a second bariatric procedure for a complications during the 6 months follow-up.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
plasma leves of oxytocin | 6 months
  Correlation between plasma leves of oxytocin (pcgr/ml) and weight loss (BMI Kg/m2) 6 months after sleeve gastrectomy

SECONDARY OUTCOMES:
sleeve gastrectomy | 6 months
  Correlation between weight 6 months after sleeve gastrectomy and fibrosis within adipose tissue

CONTACTS AND LOCATIONS:
Overall Officials: Iannelli Antonio, PhD, Principal Investigator — CHU de Nice, Service de Chirurgie
Locations (1):
- CHU de Nice, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: No